CLINICAL TRIAL: NCT07115199
Title: Remote Patient Monitoring for Chronic Hypertension During Pregnancy (REACH)
Acronym: REACH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Emily B. Rosenfeld, DO, Maternal-Fetal Medicine Faculty, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2025001233; K12TR004788 (NIH)
Record Dates: First submitted 2025-07-29; First posted 2025-08-11 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hypertension in Pregnancy
Keywords: Chronic hypertension in pregnancy; Remote Patient Monitoring
MeSH Terms: interventions — Remote Patient Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Patient monitoring (Experimental): The patients randomized to this intervention will get set up with remote patient monitoring. For these patients, blood pressure management and medication adjustment will be based on remote blood pressure measurements.
  Interventions: Procedure: Remote Patient Monitoring
- Usual Care (No Intervention): For these patients, blood pressure medication will be managed based on in office blood pressure readings.

INTERVENTIONS:
Procedure: Remote Patient Monitoring — The patients randomized to this intervention will get set up with remote patient monitoring. For these patients, blood pressure management and medication adjustment will be based on remote blood pressure measurements.
  Arms: Remote Patient monitoring

SUMMARY:
We hypothesize that frequent remote monitoring of blood pressure and real-time antihypertensive medication titration will optimize pregnancy outcomes in a clinically meaningful and cost-effective manner compared to the current standard of care. Therefore, this pilot study, as part of the K12 training support, will evaluate the feasibility of a randomized clinical trial to treat mild chronic hypertension with medication therapy to a blood pressure goal of less than 140/90 mmHg based on remote daily patient monitoring compared to in-office blood pressure readings.

DETAILED DESCRIPTION:
Hypotheses / Research Question(s) Specific Aim 1: To evaluate whether remote patient blood pressure monitoring during the antepartum period for patients with chronic hypertension will improve composite perinatal outcomes. Hypothesis: In patients with chronic hypertension, tight blood pressure control with remote patient monitoring will improve composite outcomes. Participants in the two trial arms will be compared for the frequency of composite perinatal outcomes (perinatal death, placental abruption, superimposed preeclampsia with severe features, or indicated preterm birth <35 weeks). Compliance with the assigned study group will also be assessed.

Specific Aim 2: Assess the impact of remote patient monitoring for chronic hypertension during pregnancy on changes in cardiac strain. Hypothesis: Tight blood pressure control using remote patient monitoring will decrease maladaptive cardiac remodeling during late gestation, which will persist into the postpartum period. Cardiac strain will be assessed using speckle-tracking echocardiography at enrollment and 34 to 36 weeks of gestation.

Exploratory Aim: To compare the accuracy of OB/GYN-derived Point of Care Ultrasound (POCUS) cardiac strain assessments and diastolic parameters to the echocardiogram-derived assessment, we will seek to determine if POCUS images obtained by a physician without echocardiogram training will produce reliable results compared to those obtained with an echocardiogram.

Research Significance Chronic hypertension is defined as preexisting hypertension (>=140/90 mmHg) diagnosed before 20 weeks' gestation.1 In the United States, 2-6% of all pregnancies are complicated by chronic hypertension, resulting in up to 260,000 births to women with chronic hypertension each year.1-3 There is an increasing number of patients with chronic hypertension during pregnancy,4 and chronic hypertension disproportionally impacts Black pregnant women compared to their White counterparts.5 Of those with chronic hypertension, 25-30% will develop superimposed preeclampsia with severe features.1 Additional adverse outcomes for chronic hypertension in pregnancy are substantial and include small for gestational age birth, abruption, preterm birth, and perinatal death.1,6 Chronic hypertension in pregnancy is associated with an increased risk of superimposed preeclampsia (incidence 25-30%, relative risk compared to no chronic hypertension 3-4),2,7-10 placental abruption (incidence 1.5%, relative risk 2-3),1,2,10 preterm birth before 35 weeks (incidence 18-22%, relative risk 3-4),1,3,7,9,11 and perinatal death (incidence 6-8%, relative risk 3-5).1,2,10 Recently, Tita et al.6 published the Chronic Hypertension and Pregnancy (CHAP) randomized trial of 2,408 pregnant patients with chronic hypertension. This trial showed a 21% decrease in preeclampsia by targeting a blood pressure goal of less than 140/90 mmHg. This study was conducted using in-office blood pressure measurements to titrate medication.6 Whether using home blood pressure readings to optimize treatment further improves clinical outcomes is unknown. Of the patients in the active treatment arm (n=1170), 30.2% had one of the composite primary outcomes compared to 37.0% in the control arm (n=1155). More specifically, preeclampsia with severe features occurred in 23.3%, medically indicated preterm birth before 35 weeks occurred in 12.2%, placental abruption occurred in 1.7%, and fetal or neonatal death before 28 days of life occurred in 3.5%.6 Despite the clinically meaningful reduction in the primary outcome of the CHAP trial, it is unknown if remote patient monitoring can further decrease these adverse maternal and neonatal outcomes.

With the growth of remote clinical monitoring, many patients with chronic hypertension take their blood pressure outside of a medical setting. The United States Preventive Services Task Force recommends confirmation of hypertension outside of pregnancy based on out-of-office blood pressure measurements.1 The decision to treat hypertension based on out-of-office blood pressure measurements is complicated by the fact that studies have shown that non-pregnant patients have home blood pressure measurements that are 5-15 mmHg lower than in-office readings.13 Nevertheless, studies in nonpregnant patients have shown improved blood pressure control with 12 months of remote patient monitoring versus standard treatment alone (72% versus 57%).14 If treating in-office blood pressure readings alone, it may lead to overtreatment in some patients and missed opportunities for medication titration in others.

It is unknown whether remote patient monitoring with a validated blood pressure target and medication titration protocol can further improve outcomes during pregnancy. It is also unknown if home blood pressure readings differ from in-office blood pressures, similar to nonpregnant patients. Previous studies have not shown the benefits of home blood pressure monitoring, but they lack a standardized treatment protocol and depend on individual physician judgment when making medication adjustments.15 In a randomized trial of 850 patients with hypertension, a few of whom had chronic hypertension (n=54), the authors showed a trend toward more preeclampsia diagnoses and frequent induction of labor in those with increased monitoring.16 In more than half of the patients without preexisting hypertension, elevated blood pressures were noted a month before the diagnosis of hypertension using this passive approach to monitoring.17 Notably, this study was performed before the publication of CHAP and lacked the rigorous protocol for blood pressure medication titration that is now available. To our knowledge, there has been no randomized trial of remote patient monitoring versus standard-of-care for treating mild chronic hypertension (>=140/90 mmHg) during pregnancy.

Speckle tracking echocardiography evaluates the cardiac chamber for thickening or shortening by placing myocardial speckles and tracking the motion of the cardiac chamber.18,19 Naqvi et al. have published cardiac strain outcomes in 45 healthy patients throughout pregnancy. They found that during the third trimester, the strain of all cardiac chambers decreased, and normal values for patients were published in each trimester. In these healthy pregnant individuals, an increase in intraventricular wall thickness, left ventricular mass, and left ventricular end-diastolic diameter was also noted.20 There has been limited speck tracking performed on patients with hypertensive disorders in pregnancy. A study of 85 preeclamptic patients found an increased left atrial volume index compared to normotensive patients.21 In non-pregnant patients, it has been shown to predict cardiovascular outcomes. Global peak atrial longitudinal strain assessed by speckle tracking has been shown to predict cardiovascular events (area under the receiver operator characteristic curve 0.83).22,23 By evaluating cardiac strain, we can determine if interventions during pregnancy have a protective cardiovascular effect.

Historically, most studies of antihypertensive medications have focused on treatment based on office blood pressure measurements. However, growing evidence shows that pregnant patients benefit from more frequent monitoring. A recent study showed improved pregnancy outcomes for diabetic pregnant patients (n=533) when remote patient monitoring of glucose control was implemented.24 I hypothesize that frequent remote monitoring of blood pressure and real-time antihypertensive medication titration will optimize pregnancy outcomes in a clinically meaningful and cost-effective manner compared to the current standard of care. Therefore, this pilot study, as part of the K12 training support, will evaluate the feasibility of a randomized clinical trial to treat mild chronic hypertension with medication therapy to a blood pressure goal of less than 140/90 mmHg based on remote daily patient monitoring compared to in-office blood pressure readings (Figure 1). For this trial, patients before 20 weeks' gestation will be recruited (N=50) to the remote monitoring arm (n=25) or the in-office arm (n=25). CHAP guidelines will be used to titrate medication use in each arm.

Specific Aim 1: To evaluate whether remote patient blood pressure monitoring during the antepartum period for patients with chronic hypertension will improve composite perinatal outcomes. Hypothesis: In patients with chronic hypertension, tight blood pressure control with remote patient monitoring will improve composite outcomes. Participants in the two trial arms will be compared for the frequency of composite perinatal outcomes (perinatal death, placental abruption, superimposed preeclampsia with severe features, or indicated preterm birth <35 weeks). Compliance with the assigned study group will also be assessed.

Specific Aim 2: Assess the impact of remote patient monitoring for chronic hypertension during pregnancy on changes in cardiac strain. Hypothesis: Tight blood pressure control using remote patient monitoring will decrease maladaptive cardiac remodeling during late gestation, which will persist into the postpartum period. Cardiac strain will be assessed using speckle-tracking echocardiography at enrollment and 34 to 36 weeks of gestation.

Exploratory Aim: To compare the accuracy of OB/GYN-derived Point of Care Ultrasound (POCUS) cardiac strain assessments and diastolic parameters to the echocardiogram-derived assessment, we will seek to determine if POCUS images obtained by a physician without echocardiogram training will produce reliable results compared to those obtained with an echocardiogram.

Completing this feasibility study and planned training will provide the requisite preliminary data, knowledge, and skills to apply for an R01 grant from NICHD/NHLBI during the second year of the K12. The structured research training and mentoring enabled by the K12 will substantially accelerate my transition to an independently funded physician-scientist committed to improving perinatal clinical outcomes for patients.

1.3 Research Design and Methods A. Research Procedures The pilot study aims to evaluate the feasibility of a randomized clinical trial to treat chronic hypertension with antihypertensive therapy to a blood pressure goal of less than 140/90 mm Hg based on remote patient monitoring compared to in-office blood pressure readings. The primary clinical outcome is a composite perinatal outcome (perinatal death, placental abruption, superimposed preeclampsia with severe features, or indicated preterm birth <35 weeks). Feasibility outcomes will focus on developing recruitment procedures, determining consent rate, developing and testing approaches to measure outcomes, testing blood pressure regimen, and determining the feasibility of echocardiogram assessments. One hundred patients will be enrolled from Rutgers Robert Wood Johnson University Hospital, New Brunswick, NJ.

Inclusion and exclusion criteria: Patients with a viable pregnancy <23 weeks of gestation will be screened for chronic hypertension by either identifying those currently receiving treatment for hypertensive disorders or patients with newly diagnosed or untreated chronic hypertension defined as systolic blood pressure >=140 mm Hg or diastolic blood pressure >=90 mm Hg prior to 20 weeks gestation. Patients must be 18 years of age or older and speak English or Spanish. They also must be able to sign a consent. Patients will be excluded if they have a known secondary cause of hypertension, known major fetal anomaly, known fetal demise, suspected fetal growth restriction, membrane rupture, planned termination, plan to deliver outside of the RWJ Barnabas Health system, known sensitivity to labetalol or nifedipine or unlikely to follow up in the opinion of the study staff.

Baseline assessment: Standard of care labs will be collected for all patients who have not previously had them drawn, including complete blood count, comprehensive metabolic panel, and hemoglobin A1c. An EKG is also part of the standard of care for patients with chronic hypertension in pregnancy.

Intervention: Patients will be randomized to blood pressure management based on home or in-office readings. Patients randomized to the home blood pressure arm will be supplied with a Bluetooth-enabled blood pressure monitor that interfaces with the RWJ Barnabas electronic medical record, and staff will be assigned to assess this data daily. As part of the standard of care, patients in the office blood pressure arm will be allowed to take home blood pressure readings at the discretion of their obstetrician, and that information will be recorded, but not with real-time, Bluetooth-enabled machines.

Our site previously enrolled patients in the CHAP trial, where the study Principal Investigator managed blood pressure medication. Our colleagues have agreed to let the study team manage antihypertensive medications for any patients enrolled in the REACH study.

Outcomes: Maternal and neonatal outcome data will be ascertained from medical records and recorded in RedCap. Participants in the two trial arms will be compared for the frequency of composite perinatal outcomes (perinatal death, placental abruption, superimposed preeclampsia with severe features, or indicated preterm birth <35 weeks). Cardiac strain assessments will also be collected at baseline and at 34 to 36 weeks of gestation. Finally, compliance and similarity between in-office and home blood pressure readings will be evaluated.

Specific Aim 1: I will evaluate whether remote patient blood pressure monitoring during pregnancy for patients with chronic hypertension will improve composite perinatal outcomes. The composite outcomes will include perinatal death, placental abruption, superimposed preeclampsia with severe features, or indicated preterm birth <35 weeks.

Randomization to treatment arms: Patients diagnosed with chronic hypertension will be approached at prenatal care visits and consented to the study. REDCap will be used to randomize patients in a 1:1 ratio to either in-office blood pressure or titration based on home blood pressure readings. Patients randomized to the remote patient monitoring system will be set up with a Bluetooth-enabled tablet and blood pressure cuff through the HRS system synced with electronic medical records. These patients will be instructed to take their blood pressure twice a day. Patients randomized to in-office blood pressure monitoring are still allowed to take their blood pressure at home, but no medication adjustments will be made based on home blood pressure readings. Medication adjustments in the in-office blood pressure titration arm will occur at regular intervals: every 1-4 weeks from enrollment to 28 weeks, then every 1-2 weeks from 32-40 weeks. In the remote patient monitoring arm, prenatal care visits will occur at the same interval.

Blood pressure measurements: All patients on the remote patient monitoring arm will watch an instructional video on proper ascertainment of blood pressure and will be observed taking a practice blood pressure at the time of enrollment. Instructions will follow American Heart Association guidelines13: avoid smoking, caffeinated beverages, or exercise within 30 minutes, ensure ≥5 minutes of quiet rest before blood pressure measurements, sit with back straight and supported, sit with feet flat on the floor, keep arm supported with the upper arm at heart level, and bottom of the cuff placed directly above the antecubital fossa. Two readings should be taken at least one minute apart before morning medication and in the evening before dinner. In-office blood pressures will be recorded by trained study personnel using similar requirements. All blood pressure machines will be calibrated. The feasibility and acceptability of remote patient monitoring will be evaluated.

Medication initiation and titration: If patients are currently on antihypertensive medication at the start of the study, they will continue their current medication. Antihypertensive medication will be started for patients not on medication at the time of enrollment but with mild-range blood pressures (≥140/90 mmHg) as recommended by the CHAP trial.6 Patients randomized to in-office assessment will have their blood pressure measured with an automatic cuff during their prenatal care visit. If it is ≥140/90 mmHg, the blood pressure will be repeated 5 minutes later. For blood pressure persistently above ≥140/90 mmHg, medication is increased. If a patient on the study's remote blood pressure monitoring arm has two or more blood pressures ≥140/90 mmHg within 48 hours, then blood pressure medication will be increased.

Medication selection: Either first-line medication (labetalol or nifedipine extended-release [ER]) may be initiated based on patient history or provider preference.

Labetalol will be started at 200 mg BID and increased by increments of 200 mg BID (maximum dose 2400 mg/day). Doses can be divided into TID dosing for symptoms suggesting intolerance, including headaches, fatigue, hypotension with high doses, or uncontrolled hypertension. If a patient is on TID dosing, then medication should be titrated by 100 mg TID.

Nifedipine 30 mg ER should be the initial dose, which will be increased by 30 mg ER. The maximum dose of nifedipine ER is 120 mg/day. If the maximum tolerated dose of one medication is reached, a second medication should be added.

Other medications: If a patient is enrolled in the study while taking another medication, such as metoprolol or amlodipine, that medication can be continued. For patients on methyl-dopa, we recommend switching to another more common medication, given the difficulty of obtaining methyldopa in the United States.

Frequency of blood pressure measurements:

Remote patient monitoring arm: Patients will be instructed to obtain their blood pressure with the remote monitoring system twice a day. If a patient does not take their blood pressure for 48 hours, they will be called and reminded to take their BP.

In office blood pressure arm: blood pressure will be assessed at regular office visits at the frequency described above.

Specific Aim 2: I will assess the impact of remote patient monitoring for chronic hypertension during pregnancy on changes in cardiac strain. To this end, cardiac strain assessments will be performed in a select subset of patients. Budgetary constraints will limit the number of patients, but they will be enrolled sequentially up to the maximum number allowed by the budget. Speckle-tracking echocardiography will be used to assess left ventricular strain, which can predict future deleterious outcomes.

To assess cardiac strain, speckle-tracking echocardiography will be performed at enrollment and again between 34 and 36 weeks of gestation to assess cardiac strain. This gestational age range was chosen since it is after peak volume status is reached during pregnancy.26 However, if impending preterm delivery is likely (i.e., diagnosis of superimposed preeclampsia with severe features), the assessment will be performed earlier. The information collected in this aim will be used to evaluate whether it is feasible to monitor cardiac strain with speckle tracking and analyze cardiac outcomes for pregnant people with chronic hypertension.

Exploratory Aim: This exploratory aim will investigate if POCUS cardiac strain assessments for speckle tracking can result in outcomes similar to those of an echocardiogram obtained by a trained technician. For this aim, Dr. Partho Sengupta, MD, has offered a POCUS machine and will train me to get the proper images. I will obtain POCUS cardiac images within one week of the official echocardiogram. The results of the POCUS strain study will be compared to the speckle tracking performed on the echocardiogram. We will analyze whether POCUS is a feasible alternative to more costly echocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients with a viable pregnancy <23 weeks of gestation
* Chronic hypertension is defined as: 1) Currently receiving treatment for hypertensive disorders OR 2) Newly diagnosed or untreated chronic hypertension is defined as systolic blood pressure >=140 mm Hg or diastolic blood pressure >=90 mm Hg prior to 20 weeks of gestation
* Viable pregnancy <23 weeks of gestation
* Ability to follow directions
* Ability to consent
* Speak English or Spanish

Exclusion Criteria:

* Known secondary cause of hypertension
* Known major fetal anomaly
* Known fetal demise
* Suspected fetal growth restriction
* Membrane rupture
* Planned termination
* Plan to deliver outside of the RWJ Barnabas Health system
* Known sensitivity to labetalol or nifedipine
* Unlikely to follow up, in the opinion of the study staff.
* Any medical condition that the providers feel is a contraindication to the REACH algorithm.
* Unwillingness to take blood pressure at home

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite perinatal outcomes | Delivery until 28 days after birth
  This study will examine a primary composite of perinatal outcomes (Perinatal death, placental abruption, superimposed preeclampsia with severe features, or indicated preterm birth <35 weeks)

SECONDARY OUTCOMES:
Cardiac strain | 36 weeks gestation
  Cardiac strain assessments will also be collected at baseline and at 34 to 36 weeks of gestation.
POCUS | 36 weeks gestation
  Accuracy of POCUS assessment for cardiac strain compared to echocardiograms obtained by a certified echocardiogram technologist.

OTHER OUTCOMES:
Accuracy of BP reading | From randomization to delivery (up to 36 weeks)
  Compliance and similarity between in-office and home blood pressure readings will be evaluated.
Feasibility of study procedures | From randomization to delivery (up to 36 weeks)
  Feasibility outcomes will focus on developing recruitment procedures, determining consent rate, developing and testing approaches to measure outcomes, testing blood pressure regimen, and determining the feasibility of echocardiogram assessments

CONTACTS AND LOCATIONS:
Overall Officials: Emily B Rosenfeld, DO, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenfeld EB, Sagaram D, Lee R, Sadural E, Miller RC, Lin R, Jenkins D, Blackledge K, Nikodijevic I, Rizzo A, Martinez V, Daggett EE, McGeough O, Ananth CV, Rosen T. Management of Postpartum Preeclampsia and Hypertensive Disorders (MOPP): Postpartum Tight vs Standard Blood Pressure Control. JACC Adv. 2025 Mar;4(3):101617. doi: 10.1016/j.jacadv.2025.101617. Epub 2025 Jan 31. PMID 39983612
- [Background] Kantorowska A, Cohen K, Oberlander M, Jaysing AR, Akerman MB, Wise AM, Mann DM, Testa PA, Chavez MR, Vintzileos AM, Heo HJ. Remote patient monitoring for management of diabetes mellitus in pregnancy is associated with improved maternal and neonatal outcomes. Am J Obstet Gynecol. 2023 Jun;228(6):726.e1-726.e11. doi: 10.1016/j.ajog.2023.02.015. Epub 2023 Feb 24. PMID 36841348
- [Background] Roos CJ, Auger D, Djaberi R, de Koning EJ, Rabelink TJ, Pereira AM, Bax JJ, Delgado V, Jukema JW, Scholte AJ. Relationship between left ventricular diastolic function and arterial stiffness in asymptomatic patients with diabetes mellitus. Int J Cardiovasc Imaging. 2013 Mar;29(3):609-16. doi: 10.1007/s10554-012-0129-y. Epub 2012 Sep 28. PMID 23053856
- [Background] Cameli M, Lisi M, Focardi M, Reccia R, Natali BM, Sparla S, Mondillo S. Left atrial deformation analysis by speckle tracking echocardiography for prediction of cardiovascular outcomes. Am J Cardiol. 2012 Jul 15;110(2):264-9. doi: 10.1016/j.amjcard.2012.03.022. Epub 2012 Apr 10. PMID 22497676
- [Background] Cong J, Fan T, Yang X, Shen J, Cheng G, Zhang Z. Maternal cardiac remodeling and dysfunction in preeclampsia: a three-dimensional speckle-tracking echocardiography study. Int J Cardiovasc Imaging. 2015 Oct;31(7):1361-8. doi: 10.1007/s10554-015-0694-y. Epub 2015 Jun 16. PMID 26077816
- [Background] Naqvi TZ, Meena Narayanan, Rafie R, Qamruddin S, Lee MS, Girardo ME, Daneshvar S, Wen S, Stek AM, Elkayam U. Cardiovascular Adaptation in Normal Pregnancy With 2D and 3D Echocardiography, Speckle Tracking, and Radial Artery Tonometry. JACC Adv. 2024 Nov 7;3(11):101360. doi: 10.1016/j.jacadv.2024.101360. eCollection 2024 Nov. PMID 39553379
- [Background] Heimdal A, Stoylen A, Torp H, Skjaerpe T. Real-time strain rate imaging of the left ventricle by ultrasound. J Am Soc Echocardiogr. 1998 Nov;11(11):1013-9. doi: 10.1016/s0894-7317(98)70151-8. PMID 9812093
- [Background] Blessberger H, Binder T. NON-invasive imaging: Two dimensional speckle tracking echocardiography: basic principles. Heart. 2010 May;96(9):716-22. doi: 10.1136/hrt.2007.141002. No abstract available. PMID 20424157
- [Background] Tucker KL, Hinton L, Green M, Chappell LC, McManus RJ. Using self-monitoring to detect and manage raised blood pressure and pre-eclampsia during pregnancy: the BUMP research programme and its impact. Hypertens Res. 2024 Mar;47(3):714-720. doi: 10.1038/s41440-023-01474-w. Epub 2023 Dec 7. PMID 38062200
- [Background] Chappell LC, Tucker KL, Galal U, Yu LM, Campbell H, Rivero-Arias O, Allen J, Band R, Chisholm A, Crawford C, Dougall G, Engonidou L, Franssen M, Green M, Greenfield S, Hinton L, Hodgkinson J, Lavallee L, Leeson P, McCourt C, Mackillop L, Sandall J, Santos M, Tarassenko L, Velardo C, Wilson H, Yardley L, McManus RJ; BUMP 2 Investigators. Effect of Self-monitoring of Blood Pressure on Blood Pressure Control in Pregnant Individuals With Chronic or Gestational Hypertension: The BUMP 2 Randomized Clinical Trial. JAMA. 2022 May 3;327(17):1666-1678. doi: 10.1001/jama.2022.4726. PMID 35503345
- [Background] Ashworth DC, Maule SP, Stewart F, Nathan HL, Shennan AH, Chappell LC. Setting and techniques for monitoring blood pressure during pregnancy. Cochrane Database Syst Rev. 2020 Jul 23;8(8):CD012739. doi: 10.1002/14651858.CD012739.pub2. PMID 32748394
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Groen SE, Kadrmas HM, Kerby TJ, Klotzle KJ, Maciosek MV, Michels RD, O'Connor PJ, Pritchard RA, Sekenski JL, Sperl-Hillen JM, Trower NK. Effect of home blood pressure telemonitoring and pharmacist management on blood pressure control: a cluster randomized clinical trial. JAMA. 2013 Jul 3;310(1):46-56. doi: 10.1001/jama.2013.6549. PMID 23821088
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] US Preventive Services Task Force; Krist AH, Davidson KW, Mangione CM, Cabana M, Caughey AB, Davis EM, Donahue KE, Doubeni CA, Kubik M, Li L, Ogedegbe G, Pbert L, Silverstein M, Stevermer J, Tseng CW, Wong JB. Screening for Hypertension in Adults: US Preventive Services Task Force Reaffirmation Recommendation Statement. JAMA. 2021 Apr 27;325(16):1650-1656. doi: 10.1001/jama.2021.4987. PMID 33904861
- [Background] Ray JG, Vermeulen MJ, Burrows EA, Burrows RF. Use of antihypertensive medications in pregnancy and the risk of adverse perinatal outcomes: McMaster Outcome Study of Hypertension In Pregnancy 2 (MOS HIP 2). BMC Pregnancy Childbirth. 2001;1(1):6. doi: 10.1186/1471-2393-1-6. PMID 11737873
- [Background] Livingston JC, Maxwell BD, Sibai BM. Chronic hypertension in pregnancy. Minerva Ginecol. 2003 Feb;55(1):1-13. PMID 12598838
- [Background] Powrie RO. A 30-year-old woman with chronic hypertension trying to conceive. JAMA. 2007 Oct 3;298(13):1548-58. doi: 10.1001/jama.298.13.1548. PMID 17911500
- [Background] Sibai BM, Lindheimer M, Hauth J, Caritis S, VanDorsten P, Klebanoff M, MacPherson C, Landon M, Miodovnik M, Paul R, Meis P, Dombrowski M. Risk factors for preeclampsia, abruptio placentae, and adverse neonatal outcomes among women with chronic hypertension. National Institute of Child Health and Human Development Network of Maternal-Fetal Medicine Units. N Engl J Med. 1998 Sep 3;339(10):667-71. doi: 10.1056/NEJM199809033391004. No abstract available. PMID 9725924
- [Background] Mulrow CD, Chiquette E, Ferrer RL, Sibai BM, Stevens KR, Harris M, Montgomery KA, Stamm K. Management of chronic hypertension during pregnancy. Evid Rep Technol Assess (Summ). 2000 Aug;(14):1-4. No abstract available. PMID 11019692
- [Background] Tita AT, Szychowski JM, Boggess K, Dugoff L, Sibai B, Lawrence K, Hughes BL, Bell J, Aagaard K, Edwards RK, Gibson K, Haas DM, Plante L, Metz T, Casey B, Esplin S, Longo S, Hoffman M, Saade GR, Hoppe KK, Foroutan J, Tuuli M, Owens MY, Simhan HN, Frey H, Rosen T, Palatnik A, Baker S, August P, Reddy UM, Kinzler W, Su E, Krishna I, Nguyen N, Norton ME, Skupski D, El-Sayed YY, Ogunyemi D, Galis ZS, Harper L, Ambalavanan N, Geller NL, Oparil S, Cutter GR, Andrews WW; Chronic Hypertension and Pregnancy (CHAP) Trial Consortium. Treatment for Mild Chronic Hypertension during Pregnancy. N Engl J Med. 2022 May 12;386(19):1781-1792. doi: 10.1056/NEJMoa2201295. Epub 2022 Apr 2. PMID 35363951
- [Background] Ford ND, Cox S, Ko JY, Ouyang L, Romero L, Colarusso T, Ferre CD, Kroelinger CD, Hayes DK, Barfield WD. Hypertensive Disorders in Pregnancy and Mortality at Delivery Hospitalization - United States, 2017-2019. MMWR Morb Mortal Wkly Rep. 2022 Apr 29;71(17):585-591. doi: 10.15585/mmwr.mm7117a1. PMID 35482575
- [Background] Ananth CV, Duzyj CM, Yadava S, Schwebel M, Tita ATN, Joseph KS. Changes in the Prevalence of Chronic Hypertension in Pregnancy, United States, 1970 to 2010. Hypertension. 2019 Nov;74(5):1089-1095. doi: 10.1161/HYPERTENSIONAHA.119.12968. Epub 2019 Sep 9. PMID 31495278
- [Background] Meis PJ, Goldenberg RL, Mercer BM, Iams JD, Moawad AH, Miodovnik M, Menard MK, Caritis SN, Thurnau GR, Bottoms SF, Das A, Roberts JM, McNellis D. The preterm prediction study: risk factors for indicated preterm births. Maternal-Fetal Medicine Units Network of the National Institute of Child Health and Human Development. Am J Obstet Gynecol. 1998 Mar;178(3):562-7. doi: 10.1016/s0002-9378(98)70439-9. PMID 9539527
- [Background] ACOG Practice Bulletin No. 203 Summary: Chronic Hypertension in Pregnancy. Obstet Gynecol. 2019 Jan;133(1):215-219. doi: 10.1097/AOG.0000000000003021. PMID 30575669
- [Background] Sibai BM. Chronic hypertension in pregnancy. Obstet Gynecol. 2002 Aug;100(2):369-77. doi: 10.1016/s0029-7844(02)02128-2. PMID 12151166